CLINICAL TRIAL: NCT00381147
Title: Phase III, Randomized, Double Blind Study of Low Dose Long Term Clarithromycin Versus Placebo in Treatment of Chronic Pulmonary Lesions Due to Sulfur Mustard
Brief Title: Use of Clarithromycin in Mustard-Induced Bronchiolitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baqiyatallah Medical Sciences University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S-340-14-6-1-PU-11
Record Dates: First submitted 2006-09-26; First posted 2006-09-27 (Estimated); Last update posted 2009-01-07 (Estimated); Status verified 2006-09

CONDITIONS: Bronchiolitis Obliterans; Acute Obliterating Bronchiolitis
MeSH Terms: conditions — Bronchiolitis Obliterans | interventions — Clarithromycin

INTERVENTIONS:
Drug: Clarithromycin

SUMMARY:
We looked for the effectiveness of low-dose long-term prescription of clarithromycin in mustard-induced chronic pulmonary lesions, especially bronchiolitis obliterans

ELIGIBILITY:
Inclusion Criteria:

* His/her own will to participate
* Documented chemical exposure
* Clinical, spirometric and radiological findings were compatible with BO on High Resolution Computed Tomography (HRCT)

Exclusion Criteria:

* any drug reactions during the trial
* history of sensitivity to macrolides
* diarrhea, gray stool, jaundice, eosinophilia, acute cholestatic hepatitis, pruritis, dark urine, abdominal pain, osteomatosis, depression, taste change, behavioural changes, early fatigue, odynophagia, glossitis , dizziness
* co-adminstration of: terfenadine, theophylline, carbamazepine, ergotamine, dihydroergotamine, warfarin, cisapride, digoxin, triazolam, phenytoin, steroids, any immunosuppressive, any systemic antibiotics
* using drugs that he/she cannot discontinue
* using drugs with potential interaction
* subject will to exit from the trial
* history of lobe resection of lung
* history of exacerbation in the last month prior to the beginning of trial
* continuous need to oxygen
* use of corticosteroids in last week prior to the trial beginning
* Radiographic evidence of pneumonia, active tuberculosis, lung carcinoma, or an infection that necessitated the use of an antibiotic
* exacerbating of subjects
* creatinine srum level more than normal
* increasing ALT, AST levels
* total bilirubin more twice than normal
* subjects who did not use their drugs properly

Sex: Male
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Ghanei, Professor, Study Director — Research Center of Chemical Injuries, Baqyatallah Medical Sciences University, Tehran, Iran
Locations (1):
- Baqiyatallah Medical Sciences University, Tehran, Tehran Province, Iran